CLINICAL TRIAL: NCT06347419
Title: Examining the Relationship Between Body Awareness and Spinal Stability in Individuals With Scoliosis
Brief Title: Body Awareness and Spinal Stability in Scoliosis
Status: Not yet recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İnci Hazal Ayas, Principal Investigator, Gazi University
Other Study IDs: Iayas8
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Scoliosis Idiopathic
Keywords: Body Awareness; Spinal Stability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Idiopathic scoliosis: The study group for this research comprises patients diagnosed with idiopathic scoliosis, a condition characterized by abnormal lateral curvature of the spine of unknown cause.
  Interventions: Other: Physiotherapy evaluation

INTERVENTIONS:
Other: Physiotherapy evaluation — In the physiotherapy evaluation, patients' spinal stability, rotary stability, and body awareness will be assessed.

SUMMARY:
Thirty volunteer patients diagnosed with scoliosis by a specialist physician at Gazi University Hospital Orthopedics and Traumatology Department and subsequently referred to Gazi University Physiotherapy and Rehabilitation Department for exercise training will be included in the study. The lumbar Pressure Measurement Test with Stabilizer and Rotation Stability Tests will be utilized to evaluate the spinal stability of the patients. Body awareness will be assessed using the Body Awareness Survey, comprising 18 questions. All assessments will be conducted at the Orthopedic Rehabilitation Clinic within the relevant department.

The results obtained from this study will elucidate the relationship between body awareness and spinal stability in individuals with scoliosis.

DETAILED DESCRIPTION:
The data obtained from the study will be analyzed using the Statistical Package for the Social Sciences (SPSS) software (IBM Corp., Armonk, NY, USA). Results will be presented as Mean ± Standard Deviation (X ± SD), percentage (%), or median with interquartile range (IQR), depending on their distribution normality. Data conforming to a normal distribution will be compared using the Independent Samples Student's t-test, while those not conforming will be analyzed using the Mann-Whitney U test. The relationship between variables will be assessed using the Spearman Correlation Test. A significance level of p < 0.05 will be utilized to determine statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic scoliosis by an orthopedist
* The Cobb angle measured on the standard scoliosis radiograph should fall within the range of 10°-45°.

Exclusion Criteria:

* Presence of any orthopedic or neurological disease affecting trunk and extremity mobility, excluding scoliosis.
* History of previous spine or orthopedic surgery.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with idiopathic scoliosis by a specialist physician at Gazi University Hospital, Deparment of Orthopedics and Traumatology will be included in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Spinal stability | Initial examination
  Spinal stability will be assessed utilizing the Stabilizer Biofeedback Pressure device.Participants will lie on their backs on a Stabilizer Biofeedback Pressure unit connected to a manometer. The pressurized biofeedback device will be placed under the vertebrae and in the middle of the spina iliaca posterior superior (SIPS) by the physiotherapist. The valve of the manometer will be closed, and the cuff will be inflated to a pressure of 40 mm/Hg. Participants will then be instructed to perform the posterior pelvic tilt maneuver as demonstrated and maintain the position for 10 seconds. The value indicated on the manometer will be recorded. This measurement procedure will be repeated three times, and the average of these measurements will be utilized in the subsequent statistical analysis.
Rotary Stability | Initial examination
  The Rotary Stability Test is a physical assessment used to evaluate an individual's ability to stabilize the spine and pelvis during rotational movements. During the test, the individual assumes a plank position (face down, supported by the toes and forearms) while maintaining a neutral spine alignment. Then, they are instructed to lift one arm and the opposite leg simultaneously while minimizing any rotation or movement in the torso and pelvis. The test measures the individual's ability to resist rotational forces.The patient will receive 3 points if the test is successfully repeated bilaterally, 2 points if it can be performed unilaterally, 1 point if there is a loss of balance during the test, and 0 points if the test cannot be completed.
Body Awareness | Initial examination
  Body awareness will be evaluated using the Body Awareness Questionnaire comprising 18 items. Participants will be instructed to rate each question on a scale of 1 to 7.The total score to be taken from the survey can be 126 or at least 18.Higher total scores indicate greater levels of body awareness, while lower scores suggest lower levels of body awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Hazar, Professor, Principal Investigator — Gazi University
Locations (1):
- Gazi University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No